CLINICAL TRIAL: NCT04893408
Title: Postoperative and Long-term Survival in Relation to Life-expectancy After Pancreatic Surgery in Elderly Patients
Brief Title: Pancreatic Surgery in Elderly Patients
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, carsten palnaes hansen, consultant, Rigshospitalet, Denmark
Other Study IDs: RH-C-2021-1
Record Dates: First submitted 2021-05-15; First posted 2021-05-19 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2021-05

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer, surgery, old patients
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observational study

SUMMARY:
Pancreatic cancer is mainly seen among elderly subjects as more than 85 % of all patients are diagnosed after 60 years of age. Pancreatic surgery in the elderly is usually well tolerated, and the postoperative mortality has decreased and today is less than 5 % in high-volume centers. When offering an old patient pancreatic surgery for a malignant disease it is important to evaluate not only the probability that the patient may survive the operation, but also the relevance of an operation in relation to the patient's remnant life expectancy and other treatment options than surgery. This problem has not been addressed in most studies on pancreatic surgery in the elderly, in which the outcome after surgery was the end point. The endpoints of the present study are the post-operative survival and surgical complications after major pancreatic surgery in all patients operated in the study period, and the long-term survival of patients operated for adenocarcinomas. These endpoints were set from the assumption that the postoperative mortality is related to age and comorbidity, while the long-term survival is influenced by the primary disease.

DETAILED DESCRIPTION:
Study design The study is a retrospective, descriptive register study based on data from a prospectively maintained database. Data recruitment include all patients from the age of 18 with adenocarcinoma in the pancreas, papilla of vater and duodenum operated between January 1, 2010 and December 31, 2019 with a minimum of one year post-operative follow-up. Study completion date will be December 31, 2020. Patients are divided into two cohorts, patients younger than 75 years and patients 75 years and older. Moreover, data are divided into patients with malignant and non-malignant tumors. The study is reported according to the STROCSS guidelines (www.strocssguideline.com).

Study population The study includes 1,556 consecutive patients, 1,296 patients between 18 and 75 years and 260 patients aged 75 years and older. There are 1,208 patients with malignant tumours of whom 1,020 have adenocarcinoma. The remaining 348 patients have benign or no pathologic findings but were operated for pre-malignant diseases or on suspicion of a malignant tumor.

Data collection Data are collected from our prospectively maintained database of pancreatic operations, from the electronic hospital record systems Orbit and EPIC, the Danish National Pathology Data Registry, and from the National Register of Death. All Danish Nationals have a unique Central Person Registration number that enables searching of health data. Patients from the Faroe Islands and Greenland are excluded, as they are not recorded in the Danish death register.

Outcomes Relevant postoperative complications are recorded in the study and include leakage from the pancreatic, bile or gastrojejunal anastomosis, intraabdominal hemorrhage and abscess formation or other complications with severe or fatal outcome. Outcomes are defined as postoperative complications and mortality assessed during 30- and 90-days and overall survival (OS) defined as the time from surgery to death from any cause or censoring at time of last follow-up. Hospitalization is defined as postoperative stay until discharge. In-hospital mortality is defined as all deaths from time of admission until discharge. Cancer specific mortality is defined as death from adenocarcinoma after other causes are censured. Recorded years of life lost are defined as lost years compared to the expected remnant life of an age-matched standard population. The recorded years of life lost are the number of deprived years that could have been saved, if patient had not developed an event that had shortened life.

Statistics Data are presented as median and range if not otherwise stated. Categorial data are presented as numbers or percentage and are analyzed with Fisher's exact test. Non-parametric continuous data between subgroups are analyzed with the Mann-Whitney test. The Kaplan-Meier method and the cumulative incidence function with correction for competing risks are used to estimate OS and the log-rank test to examine the differences between curves. The expected years of life lost are calculated as the difference between the area under the survival curve of the reference population and the patient population. The reference population is an age and sex matched Danish standard population. A p < 0.05 is considered statistically significant. Statistical analysis is performed with GraphPad Prism software version 6.05. (GraphPad, La Jolla, CA).

Ethics The study is a descriptive study and conducted in accordance with the principles stated in the Declaration of Helsinki. No approval is required according to the Danish National Health Board. The use of register data follows the General Data Protection Regulation of the European Union and is approved by the Danish Data Protection Agency (RH -2015-07, nr. 03616) and patients' consent. Consent for using health data was obtained before operation.

ELIGIBILITY:
Inclusion Criteria:

* all patients with pancreatic resection aged 18 years and older

Exclusion Criteria:

* patients younger than 18 years

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Danish population operated for pancreatic tumors including ductal adenocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 1556 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
postoperative mortality | 1. January 2010 to 31. December 2019
  data base study
long time survival in patients operated for pancreatic cancer | 1. January 2010 to 31. December 2019
  data base study

CONTACTS AND LOCATIONS:
Overall Officials: carsten p hansen, MD, DMSc, Principal Investigator — Rigshospitalet, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer Statistics, 2021. CA Cancer J Clin. 2021 Jan;71(1):7-33. doi: 10.3322/caac.21654. Epub 2021 Jan 12. PMID 33433946
- [Background] van Roessel S, Mackay TM, Tol JAMG, van Delden OM, van Lienden KP, Nio CY, Phoa SSKS, Fockens P, van Hooft JE, Verheij J, Wilmink JW, van Gulik TM, Gouma DJ, Busch OR, Besselink MG. Impact of expanding indications on surgical and oncological outcome in 1434 consecutive pancreatoduodenectomies. HPB (Oxford). 2019 Jul;21(7):865-875. doi: 10.1016/j.hpb.2018.10.020. Epub 2018 Dec 31. PMID 30606684
- [Background] Krautz C, Nimptsch U, Weber GF, Mansky T, Grutzmann R. Effect of Hospital Volume on In-hospital Morbidity and Mortality Following Pancreatic Surgery in Germany. Ann Surg. 2018 Mar;267(3):411-417. doi: 10.1097/SLA.0000000000002248. PMID 28379871
- [Background] Grobmyer SR, Kooby D, Blumgart LH, Hochwald SN. Novel pancreaticojejunostomy with a low rate of anastomotic failure-related complications. J Am Coll Surg. 2010 Jan;210(1):54-9. doi: 10.1016/j.jamcollsurg.2009.09.020. Epub 2009 Oct 28. PMID 20123332
- [Background] Valle JW, Palmer D, Jackson R, Cox T, Neoptolemos JP, Ghaneh P, Rawcliffe CL, Bassi C, Stocken DD, Cunningham D, O'Reilly D, Goldstein D, Robinson BA, Karapetis C, Scarfe A, Lacaine F, Sand J, Izbicki JR, Mayerle J, Dervenis C, Olah A, Butturini G, Lind PA, Middleton MR, Anthoney A, Sumpter K, Carter R, Buchler MW. Optimal duration and timing of adjuvant chemotherapy after definitive surgery for ductal adenocarcinoma of the pancreas: ongoing lessons from the ESPAC-3 study. J Clin Oncol. 2014 Feb 20;32(6):504-12. doi: 10.1200/JCO.2013.50.7657. Epub 2014 Jan 13. PMID 24419109
- [Background] Neoptolemos JP, Palmer DH, Ghaneh P, Psarelli EE, Valle JW, Halloran CM, Faluyi O, O'Reilly DA, Cunningham D, Wadsley J, Darby S, Meyer T, Gillmore R, Anthoney A, Lind P, Glimelius B, Falk S, Izbicki JR, Middleton GW, Cummins S, Ross PJ, Wasan H, McDonald A, Crosby T, Ma YT, Patel K, Sherriff D, Soomal R, Borg D, Sothi S, Hammel P, Hackert T, Jackson R, Buchler MW; European Study Group for Pancreatic Cancer. Comparison of adjuvant gemcitabine and capecitabine with gemcitabine monotherapy in patients with resected pancreatic cancer (ESPAC-4): a multicentre, open-label, randomised, phase 3 trial. Lancet. 2017 Mar 11;389(10073):1011-1024. doi: 10.1016/S0140-6736(16)32409-6. Epub 2017 Jan 25. PMID 28129987
- [Background] Conroy T, Hammel P, Hebbar M, Ben Abdelghani M, Wei AC, Raoul JL, Chone L, Francois E, Artru P, Biagi JJ, Lecomte T, Assenat E, Faroux R, Ychou M, Volet J, Sauvanet A, Breysacher G, Di Fiore F, Cripps C, Kavan P, Texereau P, Bouhier-Leporrier K, Khemissa-Akouz F, Legoux JL, Juzyna B, Gourgou S, O'Callaghan CJ, Jouffroy-Zeller C, Rat P, Malka D, Castan F, Bachet JB; Canadian Cancer Trials Group and the Unicancer-GI-PRODIGE Group. FOLFIRINOX or Gemcitabine as Adjuvant Therapy for Pancreatic Cancer. N Engl J Med. 2018 Dec 20;379(25):2395-2406. doi: 10.1056/NEJMoa1809775. PMID 30575490
- [Background] Ducreux M, Cuhna AS, Caramella C, Hollebecque A, Burtin P, Goere D, Seufferlein T, Haustermans K, Van Laethem JL, Conroy T, Arnold D; ESMO Guidelines Committee. Cancer of the pancreas: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2015 Sep;26 Suppl 5:v56-68. doi: 10.1093/annonc/mdv295. No abstract available. PMID 26314780
- [Background] Kim HT. Cumulative incidence in competing risks data and competing risks regression analysis. Clin Cancer Res. 2007 Jan 15;13(2 Pt 1):559-65. doi: 10.1158/1078-0432.CCR-06-1210. PMID 17255278
- [Background] Jindal M, Zheng C, Quadri HS, Ihemelandu CU, Hong YK, Smith AK, Dudeja V, Shara NM, Johnson LB, Al-Refaie WB. Why Do Long-Distance Travelers Have Improved Pancreatectomy Outcomes? J Am Coll Surg. 2017 Aug;225(2):216-225. doi: 10.1016/j.jamcollsurg.2017.04.003. Epub 2017 Apr 14. PMID 28414114
- [Background] van der Geest LG, Besselink MG, Busch OR, de Hingh IH, van Eijck CH, Dejong CH, Lemmens VE. Elderly Patients Strongly Benefit from Centralization of Pancreatic Cancer Surgery: A Population-Based Study. Ann Surg Oncol. 2016 Jun;23(6):2002-9. doi: 10.1245/s10434-016-5089-3. Epub 2016 Jan 21. PMID 26795767
- [Background] Huang L, Jansen L, Balavarca Y, Molina-Montes E, Babaei M, van der Geest L, Lemmens V, Van Eycken L, De Schutter H, Johannesen TB, Fristrup CW, Mortensen MB, Primic-Zakelj M, Zadnik V, Becker N, Hackert T, Magi M, Cassetti T, Sassatelli R, Grutzmann R, Merkel S, Goncalves AF, Bento MJ, Hegyi P, Lakatos G, Szentesi A, Moreau M, van de Velde T, Broeks A, Sant M, Minicozzi P, Mazzaferro V, Real FX, Carrato A, Molero X, Besselink MG, Malats N, Buchler MW, Schrotz-King P, Brenner H. Resection of pancreatic cancer in Europe and USA: an international large-scale study highlighting large variations. Gut. 2019 Jan;68(1):130-139. doi: 10.1136/gutjnl-2017-314828. Epub 2017 Nov 20. PMID 29158237
- [Background] Shamali A, De'Ath HD, Jaber B, Abuawad M, Barbaro S, Hamaday Z, Abu Hilal M. Elderly patients have similar short term outcomes and five-year survival compared to younger patients after pancreaticoduodenectomy. Int J Surg. 2017 Sep;45:138-143. doi: 10.1016/j.ijsu.2017.07.106. Epub 2017 Aug 4. PMID 28782662
- [Background] Adham M, Bredt LC, Robert M, Perinel J, Lombard-Bohas C, Ponchon T, Valette PJ. Pancreatic resection in elderly patients: should it be denied? Langenbecks Arch Surg. 2014 Apr;399(4):449-59. doi: 10.1007/s00423-014-1183-9. Epub 2014 Mar 27. PMID 24671518
- [Background] Turrini O, Paye F, Bachellier P, Sauvanet A, Sa Cunha A, Le Treut YP, Adham M, Mabrut JY, Chiche L, Delpero JR; French Surgical Association (AFC). Pancreatectomy for adenocarcinoma in elderly patients: postoperative outcomes and long term results: a study of the French Surgical Association. Eur J Surg Oncol. 2013 Feb;39(2):171-8. doi: 10.1016/j.ejso.2012.08.017. Epub 2012 Sep 19. PMID 22999411
- [Background] Melis M, Marcon F, Masi A, Pinna A, Sarpel U, Miller G, Moore H, Cohen S, Berman R, Pachter HL, Newman E. The safety of a pancreaticoduodenectomy in patients older than 80 years: risk vs. benefits. HPB (Oxford). 2012 Sep;14(9):583-8. doi: 10.1111/j.1477-2574.2012.00484.x. Epub 2012 May 29. PMID 22882194
- [Background] Hatzaras I, Schmidt C, Klemanski D, Muscarella P, Melvin WS, Ellison EC, Bloomston M. Pancreatic resection in the octogenarian: a safe option for pancreatic malignancy. J Am Coll Surg. 2011 Mar;212(3):373-7. doi: 10.1016/j.jamcollsurg.2010.10.015. Epub 2011 Jan 12. PMID 21227721
- [Background] Lee MK, Dinorcia J, Reavey PL, Holden MM, Genkinger JM, Lee JA, Schrope BA, Chabot JA, Allendorf JD. Pancreaticoduodenectomy can be performed safely in patients aged 80 years and older. J Gastrointest Surg. 2010 Nov;14(11):1838-46. doi: 10.1007/s11605-010-1345-1. Epub 2010 Sep 8. PMID 20824366
- [Background] Hardacre JM, Simo K, McGee MF, Stellato TA, Schulak JA. Pancreatic resection in octogenarians. J Surg Res. 2009 Sep;156(1):129-32. doi: 10.1016/j.jss.2009.03.047. Epub 2009 May 3. PMID 19592032
- [Background] Makary MA, Winter JM, Cameron JL, Campbell KA, Chang D, Cunningham SC, Riall TS, Yeo CJ. Pancreaticoduodenectomy in the very elderly. J Gastrointest Surg. 2006 Mar;10(3):347-56. doi: 10.1016/j.gassur.2005.12.014. PMID 16504879
- [Background] Renz BW, Khalil PN, Mikhailov M, Graf S, Schiergens TS, Niess H, Boeck S, Heinemann V, Hartwig W, Werner J, Bruns CJ, Kleespies A. Pancreaticoduodenectomy for adenocarcinoma of the pancreatic head is justified in elderly patients: A Retrospective Cohort Study. Int J Surg. 2016 Apr;28:118-25. doi: 10.1016/j.ijsu.2016.02.064. Epub 2016 Feb 21. PMID 26906329
- [Background] Sultana A, Smith CT, Cunningham D, Starling N, Neoptolemos JP, Ghaneh P. Meta-analyses of chemotherapy for locally advanced and metastatic pancreatic cancer. J Clin Oncol. 2007 Jun 20;25(18):2607-15. doi: 10.1200/JCO.2006.09.2551. PMID 17577041
- [Background] Burris HA 3rd, Moore MJ, Andersen J, Green MR, Rothenberg ML, Modiano MR, Cripps MC, Portenoy RK, Storniolo AM, Tarassoff P, Nelson R, Dorr FA, Stephens CD, Von Hoff DD. Improvements in survival and clinical benefit with gemcitabine as first-line therapy for patients with advanced pancreas cancer: a randomized trial. J Clin Oncol. 1997 Jun;15(6):2403-13. doi: 10.1200/JCO.1997.15.6.2403. PMID 9196156
- [Background] Conroy T, Desseigne F, Ychou M, Bouche O, Guimbaud R, Becouarn Y, Adenis A, Raoul JL, Gourgou-Bourgade S, de la Fouchardiere C, Bennouna J, Bachet JB, Khemissa-Akouz F, Pere-Verge D, Delbaldo C, Assenat E, Chauffert B, Michel P, Montoto-Grillot C, Ducreux M; Groupe Tumeurs Digestives of Unicancer; PRODIGE Intergroup. FOLFIRINOX versus gemcitabine for metastatic pancreatic cancer. N Engl J Med. 2011 May 12;364(19):1817-25. doi: 10.1056/NEJMoa1011923. PMID 21561347
- [Background] Von Hoff DD, Ervin T, Arena FP, Chiorean EG, Infante J, Moore M, Seay T, Tjulandin SA, Ma WW, Saleh MN, Harris M, Reni M, Dowden S, Laheru D, Bahary N, Ramanathan RK, Tabernero J, Hidalgo M, Goldstein D, Van Cutsem E, Wei X, Iglesias J, Renschler MF. Increased survival in pancreatic cancer with nab-paclitaxel plus gemcitabine. N Engl J Med. 2013 Oct 31;369(18):1691-703. doi: 10.1056/NEJMoa1304369. Epub 2013 Oct 16. PMID 24131140